CLINICAL TRIAL: NCT02115672
Title: Phase I/II Study Using Imatinib and s.c. BL-8040 (Novel Anti CXCR4 Antagonist) for Improving Molecular Response in Chronic Myelogenous Leukemia (CML) Patients in First Chronic Phase Achieving Less Than Optimal Response With Imatinib.
Brief Title: Imatinib and BL-8040 (Novel Anti CXCR4 Antagonist) for Improving Molecular Response in Chronic Myelogenous Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: loss of support
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0575-AN-CTIL
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; imatinib; CXCR4 antagonist; BL-8040
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — 4-fluorobenzoyl-TN-14003

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BL-8040 (Experimental): Patients with chronic phase CML on Imatinib therapy (400 mg/day) achieving less than an optimal response will be treated with sc injections of BL-8040, while continuing Imatinib. The first part of the study will include escalating dose groups. Up to 4 dose levels will be investigated starting at dose level 1. Patients will be accrued in a conventional 3+3 design. Applying this study design, the first cohort of 3 patients will be treated at dose level 1 (0.5 mg/kg) on Day 1, 15, 29 and 43. Patients will continue taking Imatinib 400 mg/day throughout the study. Dose escalation will continue until the maximal tolerated dose (MTD) is established and protocol specific stopping rules for toxicity are met. If no MTD is reached, dose escalation will continue up to dose level 4 (1.25 mg/kg).
  Interventions: Drug: BL-8040

INTERVENTIONS:
Drug: BL-8040 — BL-8040 will be added to imatinib to improve CML response.

SUMMARY:
The aim of the study is to test the safety and efficacy of BL-8040 (a CXCR4 antagonist) in improving the response to imatinib in CML patients not achieving an optimal response with imatinib alone.

DETAILED DESCRIPTION:
To improve cytogenetic and molecular response of CML patients receiving Imatinib, who have not achieved an optimal response according to European LeukemiaNet (ELN) definitions , or MR4 after 24 months with Imatinib. This will be achieved by addition of the CXCR4 antagonist BL-8040, mobilizing CML leukemia stem cells from their protective bone marrow niche and exposing them to Imatinib and BL-8040-mediated apoptosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women subjects aged 18 to 70, inclusive.
2. Confirmed diagnosis of chronic phase CML according to the WHO criteria (WHO 2008)
3. CML patients with sub-optimal response to Tyrosine Kinase Inhibitors, defined as "warning" in the ELN recommendations:

   Following 3 months: BCR-ABL1 > 10%, and/or Ph+ 36-95% Following 6 months: BCR-ABL1 1-10%, and/or Ph + 1-35% Following 12 months: BCR-ABL1 0.1-1 % Following 24 months: Less than MR4
4. Clinical laboratory values should be as follows:

   White blood cell count < 30 X 10*9/L Creatinine < 1.5 ULN
5. Women of childbearing potential and all men must agree to use approved form of contraception
6. Subject is able and willing to comply with the requirements of the protocol.
7. Subject is able to voluntarily provide written informed consent.

Exclusion Criteria:

1. CML patients not in chronic phase.
2. CML patients receiving Tyrosine Kinase Inhibitors other than Imatinib.
3. CML patients receiving Imatinib > 400 mg/day.
4. Patients not able to sign informed consent.
5. Known allergy or hypersensitivity to any of the test compounds or materials or contraindication to test product.
6. Low Performance Status (ECOG > 2).
7. Abnormal liver function tests:

   1. Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) 2 x upper limit of normal (ULN).
   2. Serum bilirubin. Total bilirubin > 2.0 mg/dL (34 µmol/L), conjugated bilirubin > 0.8 mg/dL
8. Abnormal left ventricular ejection fraction, < 40 %.
9. Subject has concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place him/her at unacceptable risk, including, but not limited to:

   1. Subject has been diagnosed or treated for another malignancy within 3 years of enrolment, except in situ malignancy, or low-risk prostate, skin or cervix cancer after curative therapy
   2. A co-morbid condition which, in the view of the Investigators, renders the subject at high risk from treatment complications.
10. Women subjects who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of BL-8040 in combination with Imatinib in CML patients | 4 months
  The investigators will assess the safety of the BL-8040 by grading of toxicities according to standard Common Toxicity Criteria for Adverse Effects (CTCAE) criteria.

SECONDARY OUTCOMES:
To assess the clinical efficacy of BL-8040 in combination with Imatinib | 2 years
  The cytogenetic and molecular response will be assessed by standard FISH and PCR test according to established criteria.

OTHER OUTCOMES:
To assess additional pharmacodynamic parameters relevant to CXCR4 inhibition | 2 months
  The investigators will test CXCR4 receptor occupancy and expression and additional pharmacodynamic endpoints relevant to CXCR4 inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel